CLINICAL TRIAL: NCT05727189
Title: A Phase 1 Safety, Tolerability and Pharmacokinetic Study of R-Idazoxan HCl Extended-Release (TR-01-XRR), S-Idazoxan HCl Extended-Release (TR-01-XRS) and Racemic Idazoxan HCl Extended-Release (TR-01-XR) in Healthy Participants
Brief Title: A Study of Idazoxan in Healthy Participants
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Terran Biosciences Australia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TR01-XR-101
Record Dates: First submitted 2023-01-25; First posted 2023-02-14 (Actual); Last update posted 2023-11-27 (Actual); Status verified 2023-11

CONDITIONS: Healthy
MeSH Terms: interventions — Tablets

STUDY DESIGN:
Intervention Model Description: Part 1: Parallel group comparison, single dose level of 5 forms of the investigational study drug.
  Part 2: Parallel group comparison, single dose escalation (3 dose levels) of 4 forms investigational study drug and placebo.
  Part 3: Placebo controlled, multiple dose cross-over within 4 parallel group comparison.
  Part 4: Single-dose food effect cross-over.
Who Masked: Participant, Investigator
Masking Description: Part 1: Open Label Part 2: Double-blind Placebo Controlled Part 3: Double-blind Placebo Controlled Part 4: Open Label
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part 1 Single Dose (Experimental): Parallel group comparison, single dose level of 5 forms of the investigational study drug.
  Interventions: Drug: TR-01-XRR (1); Drug: TR-01-XRR (2); Drug: TR-01-XRR (3); Drug: TR-01-XRS; Drug: TR-01-XR
- Part 2: Single escalating doses (Experimental): Parallel group comparison, single p.o. dose escalation (3 dose levels) of 4 forms investigational study drug and placebo administered to two sequential cohorts. Dose Level 1 will be administered to the first cohort. Dose Levels 2 and 3 will be administered to a subsequent cohort. Dose levels in this cohort are separated by a 7-day washout period. Doses to be determined by review of data from Part 1.
  Interventions: Drug: TR-01-XRR (1); Drug: TR-01-XRS; Drug: TR-01-XR; Drug: TR-01-IR; Drug: Placebo
- Part 3: Multiple Dose (Experimental): Parallel group comparison of 4 active treatments dosed p.o. x 4 days. Each active is dosed in a 2-period placebo-controlled crossover separated by a 5-day washout. Doses to be determined by review of data from Part 2.
  Interventions: Drug: TR-01-XRR (1); Drug: TR-01-XRS; Drug: TR-01-XR; Drug: TR-01-IR; Drug: Placebo
- Part 4: Food Effects (Experimental): Two-period single p.o. dose fasted/fed crossover separated by 5-day washout period. Dose to be determined by review of data from Part 2.
  Interventions: Drug: TR-01-XRR (1)

INTERVENTIONS:
Drug: TR-01-XRR (1) — Extended-release form
  Other Names: R-Idazoxan HCL Extended Release (medium release rate) Tablet
Drug: TR-01-XRR (2) — Extended-release form
  Other Names: R-Idazoxan HCL Extended Release (faster release rate) Tablet
  Arms: Part 1 Single Dose
Drug: TR-01-XRR (3) — Extended-release form
  Other Names: R-Idazoxan HCL Extended Release (slower release rate) Tablet
  Arms: Part 1 Single Dose
Drug: TR-01-XRS — Extended-release form
  Other Names: S-Idazoxan Extended Release Tablet
  Arms: Part 1 Single Dose; Part 2: Single escalating doses; Part 3: Multiple Dose
Drug: TR-01-XR — Extended-release form
  Other Names: Racemic Idazoxan HCL Extended Release Tablet
  Arms: Part 1 Single Dose; Part 2: Single escalating doses; Part 3: Multiple Dose
Drug: TR-01-IR — Active comparator
  Other Names: Idazoxan HCL Immediate Release Tablet
  Arms: Part 2: Single escalating doses; Part 3: Multiple Dose
Drug: Placebo — Placebo comparator
  Other Names: Matching Placebo Tablet
  Arms: Part 2: Single escalating doses; Part 3: Multiple Dose

SUMMARY:
Four-part study of the safety, tolerability and pharmacokinetics of 3 forms of TR-01-XRR, 1 form of TR-01-XRS, and 1 form of TR-01-XR in healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18 and 32 kg/m2
* Medically healthy without clinically significant or relevant medical history

Exclusion Criteria:

* Evidence of recurrent disease, physical illness or medical condition that could affect action, absorption or disposition of investigational products
* Use of any prescription or over-the-counter medication that cannot be discontinued for the duration of the study
* Impaired renal function
* Cardiac abnormalities
* Positive HIV, HBsAg or HCV
* Positive test for alcohol, drugs of abuse or cotinine

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-02-14 (Actual); Primary Completion 2024-03 (Estimated); Study Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events based on clinical observation and participant report | Through study completion up to 25 days after initial dose
  Clinically observed adverse events include findings from physical examination, vital sign, ECG and laboratory assessments (hematological and clinical chemistry laboratory panels). Participant report includes any side effect reported by a participant during the study.
Area under the plasma concentration-time curve (AUC) | Up to 120 hours after dose
  To evaluate drug exposure over specified measurement time frame
Maximum plasma concentration (Cmax) | Up to 120 hours after dose
  To evaluate peak drug concentration achieved during specified measurement time frame
Time to maximum plasma concentration (Tmax) | Up to 120 hours after dose
  To evaluate time to achieve peak concentration during specified measurement time frame
Terminal elimination rate constant | Up to 120 hours after dose
  To evaluate rate of drug elimination
Terminal elimination half-life (T1/2) | Up to 120 hours after dose
  To evaluate time over which drug concentration is decreased by half
Apparent total clearance from plasma (CL/F) | Up to 120 hours after dose
  To evaluate rate of drug clearance
Apparent volume of distribution (Vz/F) | Up to 120 hours after dose
  To evaluate extent of drug distribution in the body

SECONDARY OUTCOMES:
Relative bioavailability (Frel) | Over 120 hours after dose
  To compare single dose oral bioavailability in fed and fasted states

CONTACTS AND LOCATIONS:
Overall Officials: Robert Fishman, MD, Study Director — Clinical Lead Consultant
Locations (2):
- Australia (2):
  - Scientia Clinical Research, Randwick, New South Wales
  - CMAX Clinical Research, Adelaide, South Australia

IPD SHARING:
Plan to Share IPD: No